CLINICAL TRIAL: NCT04409782
Title: Education About Health and Cancer Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Dartmouth College (Other)
Responsible Party: Principal Investigator, Judith R. Rees, Associate Professor of Epidemiology; Associate Professor of Community and Family Medicine; Associate Director for Community Outreach and Engagement, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: D20039; P30CA023108-40S4 (NIH)
Record Dates: First submitted 2020-05-15; First posted 2020-06-01 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Cancer
Keywords: Education; Clinical Trial; Research
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Our study will be largely advertised to DCC's patients and caregivers via electronic provider portal BPA. Providers will provide prospective participants with a link to an online survey where they can consent, complete eligibility screening, the pretest, and contact information.
  Interventions: Other: Electronic portal education
- Arm 2 (Experimental): People with social medial accounts (e.g. Facebook) will receive a message about the study (e.g. via a geospatially targeted Facebook ad) and have the option to enroll in the study if meeting eligibility criteria, with some participating in online follow-up.
  Interventions: Other: Online educational video

INTERVENTIONS:
Other: Electronic portal education — Participants will receive education via an electronic portal covering the key messages pertaining to cancer research studies and clinical trials. Data will be collected via pre- and post-tests. The post-test includes questions to pre-screen participants for eligibility into cancer research studies and clinical trials; as appropriate, study participants will be referred to those study/trial/clinical teams for follow-up.
  Arms: Arm 1
Other: Online educational video — Participants will receive online education via a video and written web content. Key messages will include information pertaining to cancer research studies and clinical trials. Data will be collected via pre- and post-tests. The post-test includes questions to pre-screen participants for eligibility into cancer research studies and clinical trials; as appropriate, study participants will be referred to those study/trial/clinical teams for follow-up.
  Arms: Arm 2

SUMMARY:
This study investigates different ways to educate rural residents living in New Hampshire and Vermont about cancer research studies and clinical trials to increase knowledge of, increase positive attitudes toward, and encourage enrollment in cancer research studies and clinical trials. The information learned from this study will contribute to a nation-wide initiative to educate the public about clinical trials, including a nation-wide evaluation of that initiative. The results of this study may also help researchers understand how education about clinical trials/research affects knowledge of and attitudes toward cancer research and clinical trials, as well as behavioral intentions and actual behaviors related to enrolling in cancer research studies and clinical trials.

DETAILED DESCRIPTION:
The study team will implement and evaluate the research study and clinical trials education in two experimental arms-

1. electronic portal education about clinical trials and cancer research (Aim 1a)
2. online education via an online video about clinical trials and cancer research (Aim 1b)

The education in both formats will be based on a set of key messages that cover information about research studies and clinical trials, including what research studies are, the benefits, the risks, and connection to available research studies and clinical trials

Experimental Arm 1 (Aim 1a):

Implement electronic portal education regarding what clinical trials and cancer research are and evaluate the effect on knowledge of, attitudes and behavioral intentions toward, and actual enrollment into clinical trials and cancer research studies.

We will evaluate educational outputs from electronic portal regarding what clinical trials and cancer research studies are. The educational content for videos was developed with the National Cancer Institute (NCI) toolkit as a foundation, with additional content added to adapt to our local institution, culture, and patient needs. The videos learning objectives focus on improving participants' knowledge about what clinical trials and cancer research studies are and how to access trials and studies, increase positive attitudes toward participating in trials and studies, and increase their intent to enroll in trials and studies.

Providers will receive a BPA indicating patient may qualify to participate in the education survey. See enclosed invitation language. Providers will also have the option to include After Visit Summary (AVS) to Patient Notes that will contain invitation link. Patients will receive a link to the survey. If they choose to take part in the study, they will do so by completing the online consent, eligibility screening, pre-test, and contact information before the class they are registered for; attend the class; and complete the post-test after the class to assess achievement of the learning objectives. They will also be asked a series of questions to assess their eligibility for existing DCC clinical trials and research studies.

Experimental Arm 2 (Aim 1b):

Implement online education regarding what clinical trials and cancer research are and evaluate the effect on knowledge of, attitudes and behavioral intentions toward, and actual enrollment into clinical trials and cancer research studies.

Participants will watch a video and view website materials ('online module') developed by DCC using messaging provided by the National Cancer Institute (NCI) and tailored to our local context. The online module's learning objectives will focus on improving participants' knowledge about what clinical trials and cancer research studies are and how to access trials and studies, increase positive attitudes toward participating in trials and studies, and increase their intent to enroll in trials and studies. Eligible participants will complete pre- and post- surveys to assess achievement of the learning objectives, and they will also be asked a series of questions to assess their eligibility for existing DCC clinical trials and research studies (see enclosed questions).

ELIGIBILITY:
Inclusion Criteria for Experimental Arm 1 (portal education):

- Participants will come from Dartmouth Cancer Center electronic provider portal EDH/Epic. They will receive an invitation to participate in this research study only after accessing a Qualtrics survey.

Inclusion Criteria for Experimental Arm 2 (online education):

- Participants must be a resident of one of the RUCC 7-9 counties in NH or VT: Coos, Sullivan Counties in New Hampshire, or Caledonia, Windsor, Windham, Orange, Orleans, Lamoille or Essex Counties in Vermont. They will be invited to participate in the study through social media, listservs, or from flyers in community settings.

Exclusion Criteria for both Experimental Arms:

- Cognitive impairment preventing participation in informed consent process

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2020-10-31 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Percent change in participant knowledge related to what cancer research studies and clinical trials are as assessed before and after educational intervention | Pre-test questionnaire administered before educational intervention; post-test questionnaire administered after educational intervention
  A pre-test and post-test knowledge questionnaire conducted with participants to assess any changes in knowledge related to key learning outcomes expected from the educational intervention (assessed via percent of correct and incorrect responses to 19 true/false questions and 6 multiple choice questions).
Percent change in attitudes and behavioral intentions toward enrolling in clinical trials | Pre-test questionnaire administered before educational intervention; post-test questionnaire administered after educational intervention
  A pre-test and post-test questionnaire conducted with participants to assess any changes in attitudes and behavioral intentions related to clinical trial enrollment (assessed via 4 Likert-scale questions)
Percent change in enrollment status in cancer research studies and clinical trials as measured by tracking individual enrollment statuses at the time of intervention and after education | Tracking from time of study participation in educational intervention and following study participants for six months monitoring change in enrollment status in cancer research and clinical trials
  Actual enrollment into a clinical trial or cancer research study will be assessed via Dartmouth Cancer Center (DCC) Office of Clinical Research enrollment records over 6 months post-intervention. Enrollment records for specified DCC trials/research studies will also be assessed, and change in enrollment status in cancer research or clinical trials will be measured by direct participant's active status in cancer research or clinical trials project participation.

CONTACTS AND LOCATIONS:
Overall Officials: Judith R Rees, BM, BCh, MPH, PhD, Principal Investigator — Geisel School of Medicine at Dartmouth College
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT04409782/Prot_000.pdf